CLINICAL TRIAL: NCT01045005
Title: Doppler Ultrasound Investigation of Ocular and Skeletal Microcirculations in Health and Disease
Brief Title: Doppler Ultrasound Investigation of Microcirculations
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05060CL-A
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes; Endothelial dysfunction; Doppler Ultrasound Velocity Waveforms
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Carbon Dioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Type 1 Diabetes (Active Comparator): Subjects with type 1 diabetes mellitus who are administered oxygen and carbon dioxide
  Interventions: Other: Administration of Oxygen and carbon dioxide
- Control Subjects (Active Comparator): Healthy volunteers administered oxygen and carbon dioxide via respiratory apparatus
  Interventions: Other: Administration ofOxygen and carbon dioxide

INTERVENTIONS:
Other: Administration ofOxygen and carbon dioxide — Inhalation of 100% oxygen and 4% carbon dioxide. This is non-harmful/non-toxic and will be given according to protocol previously described in the literature. It will be administered for a maximum of 4 minutes.
  Arms: Control Subjects
Other: Administration of Oxygen and carbon dioxide — Inhalation of 100% oxygen and 4% carbon dioxide. This is non-harmful/non-toxic and will be given according to protocol previously described in the literature. It will be administered for a maximum of 4 minutes.
  Arms: Type 1 Diabetes

SUMMARY:
The investigators aim to show that quantitative analysis of doppler flow velocity waveforms i.e. ultrasound which is a non-invasive and very safe means of assessing blood flow; recorded in the proximity of terminal microvascular beds of interest, (i.e. the forearm and ocular circulation) can sensitively detect and track local changes in microvascular haemodynamics i.e. the function of the small blood vessels that are found in the back of the eye and in the forearm.

The investigators also aim to relate change in the doppler spectral flow velocity waveform i.e. the ultrasound signal, in the central retinal artery to changes in geometry and tone of the vasculature (or changes in the structure and function of small blood vessels) in response to inhaled oxygen and carbon dioxide. The geometry and tone of the vasculature (or Blood Vessels) can be measured by taking photographs of the back of the eye.

DETAILED DESCRIPTION:
Diabetes mellitus significantly increases the risk for both small and large blood vessel complications e.g. diabetic eye problems and coronary heart disease. Vital organs such as the eye, kidney, heart and brain represent well- recognized preferential targets in patients with diabetes mellitus. The presence of such end-organ damage powerfully influences cardiovascular risk and the benefits of therapeutic interventions. Unfortunately, by the time symptoms develop or events occur as manifestations of target-organ damage, the disease process is already at an advanced stage. Although not traditionally viewed as an end-organ, it is altered structure and function of arterial small blood vessels that acts as the substrate for accelerated disease development and the increased occurrence of vascular events in patients with diabetes mellitus. The ability to detect and monitor sub-clinical damage, representing the cumulative and integrated influence of all risk factors in impairing arterial wall integrity, holds potential to further refine cardiovascular risk stratification and enable early intervention to prevent or attenuate disease progression.

Data derived from analysis of arterial waveforms, that marks the presence of impaired pulsatile function in the arterial system, has been shown to predict future cardiovascular risk. As consistent abnormalities in the arterial pulse wave shape have been recognized for many years in diabetic subjects there has been a growing interest in quantifying changes in the pulse contour to provide information about the status of the vasculature in diabetes. These original observations have been confirmed in more recent studies in patients with type 1 and type 2 diabetes mellitus and are detected prior to the development of clinical complications of the disease.

Analysis of the pulse contours recorded from sites in large conduit arteries identify structural and functional abnormalities predominantly in the systemic microvasculature, as small arteries and arterioles are recognised as the major sites for wave reflection that alters pulse contour morphology. It is recognised that techniques providing a global assessment of the circulation may not capture and cannot localise findings to a specific site or target-organ of interest in the arterial system. Microcirculation is a collective term for the smallest segments of the vascular system and is a major site of control of vascular resistance. It includes arterioles and capillaries and is considered to be a continuum rather than a distinct site of resistance control. Importantly, it is recognised as sites were the earliest manifestations of cardiovascular disease, especially inflammatory processes occur. The microvasculature may therefore constitute a preferential target or be primarily involved in the pathogenesis of disease and represents an important regional target for therapeutic interventions. Further, retinal photography and standardised grading provides a unique opportunity to study retinal microvascular characteristics including retinopathy and change in arteriolar (or blood vessel) structure and function. Improved methods of assessment to study the retinal microvascular network holds potential to improve prediction of risk, identify high risk groups and act as a window to monitor the effects of possible drug interventions.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for study patients must be older than 18 years.
* All patients will have undergone an extensive clinical evaluation performed at the Belfast City Hospital diabetes clinic that includes retinal photography.
* Patients will be eligible for the study if they are in stable control of their diabetes with a haemoglobin of A1c between 6.5 and 10%.
* Patients will be eligible if they have background retinopathy. The control subjects will be healthy individuals; and will be age and sex matched for the disease population.

Exclusion Criteria:

* Patients with proliferative retinopathy or those undergoing laser therapy will be excluded from study. This would make assessment of the retinal arteriolar structure very difficult.
* Patients will also be excluded if they have hypertension (a blood pressure >140/90mmHg) or taking antihypertensive drugs. The investigators know that the presence of hypertension will have an effect on the retinal waveforms and structure.
* Patients will also be excluded if they have any significant renal disease (GFR <60ml min) or a history of cardiovascular or cerebrovascular complications.
* Patients with microalbuminuria (>3 g/min) can be included in the study but would be asked to stop their medication (e.g. ACE inhibitor) for 5 days prior to the study period. It should be mentioned that the risk associated with stopping this effective medication for such a period of time is minimal. This has been common practice in our department in a number of previous studies, and in the published literature. This will be clearly communicated to the patient in the patient information sheet, in the patient consent form; and in the discussion/process of obtaining informed consent with the patient

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Doppler Blood flow velocity waveforms measured at rest and after administration of oxygen and carbon dioxide | At initial visit and then yearly

SECONDARY OUTCOMES:
Radial Artery pressure waveforms | At initial visit and then yearly

CONTACTS AND LOCATIONS:
Overall Officials: Gary E McVeigh, MD PhD FRCP, Principal Investigator — Queens University Belfast
Locations (1):
- Department of Therapeutics and Pharmacology, Queens University Belfast, Belfast, Antrim, United Kingdom

REFERENCES:
- [Background] Wright SA, O'Prey FM, Hamilton PK, Lockhart CJ, McCann A, McHenry MT, McGivern RC, Plumb R, Finch MB, Bell AL, McVeigh GE. Colour Doppler ultrasound of the ocular circulation in patients with systemic lupus erythematosus identifies altered microcirculatory haemodynamics. Lupus. 2009 Oct;18(11):950-7. doi: 10.1177/0961203309104865. PMID 19762395
- [Background] Agnew CE, Rea DJ, McCann AJ, Lockhart CJ, Hamilton PK, Quinn CE, McVeigh GE, McGivern RC. Root-MUSIC analysis of nitric oxide-mediated changes in ophthalmic artery blood flow velocity waveforms. Med Eng Phys. 2009 Sep;31(7):799-805. doi: 10.1016/j.medengphy.2009.03.003. Epub 2009 Apr 16. PMID 19375374
- [Background] Lockhart CJ, Hamilton PK, Quinn CE, McVeigh GE. End-organ dysfunction and cardiovascular outcomes: the role of the microcirculation. Clin Sci (Lond). 2009 Feb;116(3):175-90. doi: 10.1042/CS20080069. PMID 19118490
- [Background] Lockhart CJ, Hamilton PK, McVeigh KA, McVeigh GE. A cardiologist view of vascular disease in diabetes. Diabetes Obes Metab. 2008 Apr;10(4):279-92. doi: 10.1111/j.1463-1326.2007.00727.x. Epub 2007 Oct 15. PMID 17941877
- [Background] Hamilton PK, Lockhart CJ, Quinn CE, McVeigh GE. Arterial stiffness: clinical relevance, measurement and treatment. Clin Sci (Lond). 2007 Aug;113(4):157-70. doi: 10.1042/CS20070080. PMID 17623012
- [Background] Lockhart CJ, Gamble AJ, Rea D, Hughes S, McGivern RC, Wolsley C, Stevenson M, Harbinson MT, Plumb RD, McVeigh GE. Nitric oxide modulation of ophthalmic artery blood flow velocity waveform morphology in healthy volunteers. Clin Sci (Lond). 2006 Jul;111(1):47-52. doi: 10.1042/CS20050365. PMID 16499475